CLINICAL TRIAL: NCT03801681
Title: Risk Assessment of Cardiac ARrhythmias in Patients With MYocarditis
Brief Title: ARrhythmias in MYocarditis
Acronym: ARMY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Krzysztof Ozieranski, Principal Investigator, Medical University of Warsaw
Other Study IDs: ARMY
Record Dates: First submitted 2019-01-05; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Myocarditis; Heart Failure; Endomyocardial Biopsy; Arrythmia; Sudden Cardiac Death; Biomarker; Cardiomyopathy
Keywords: myocarditis; heart failure; endomyocardial biopsy; arrythmia; sudden cardiac death; biomarker; cardiomyopathy; high-sensitive troponin; galectin-3; st-2; NT-proBNP
MeSH Terms: conditions — Myocarditis; Heart Failure; Arrhythmias, Cardiac; Death, Sudden, Cardiac; Cardiomyopathies | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myocarditis: patients with clinically suspected myocarditis
  Interventions: Diagnostic Test: ECG holter monitoring

INTERVENTIONS:
Diagnostic Test: ECG holter monitoring — patients will be monitored using ECG-holter

SUMMARY:
Myocarditis promotes the occurrence of serious cardiac arrhythmias and conduction disorders which may lead to sudden cardiac death, the need for catheter ablation of arrhythmia or implantation of a cardioverter-defibrillator or pacemaker. The aim of the study is to fill the evidence gap regarding the type and burden of arrhythmias in patients with myocarditis and their correlation with clinical parameters, biomarkers and additional tests. During a multi-center observational study, patients will be subjected to prolonged ECG monitoring. As a result, a risk scale will be created that can facilitate the identification of patients with an increased risk of arrhythmia and further specifying recommendations for therapeutic management.

DETAILED DESCRIPTION:
Myocarditis is a serious social problem, usually affecting young or middle-aged people. Making of the diagnosis of myocarditis, due to the varied course of the disease, is a significant challenge, therefore clinical suspicion of myocarditis is based on symptoms and abnormalities in additional tests (ECG, echocardiography, magnetic resonance of the heart, biomarkers), which should be confirmed by cardiac biopsy. Despite the fact that in the majority of patients myocarditis occurs in a mild and uncomplicated manner, in some patients the inflammatory process progresses leading to dilated cardiomyopathy, end-stage heart failure and often to the need for heart transplantation. Myocarditis also promotes the occurrence of severe arrhythmias and conduction which may lead to sudden cardiac death (myocarditis is confirmed in autopsy even in 2-42% of cases), the need for percutaneous ablation of arrhythmia, cardioverter-defibrillator implantation or cardiac stimulator.

In order to better identify the causes and improve the diagnosis and treatment of myocarditis, new data are needed including biomarkers (including biochemical, genetic, immunohistochemical biomarkers) responsible for the process of necrosis, fibrosis, haemodynamic stress of myocardium in the course of myocarditis, as well as studies aimed at identifying pathogens that cause myocarditis and factors predisposing to the onset of myocarditis. In addition, there is no systematic information on the type and burden of arrhythmias and their variability over time. A significant deficiency of research in the field of the above biomarkers and the severity of arrhythmia in the course of myocarditis translates into the lack of clear recommendations on the myocarditis management from the scientific societies and often leads to wrong therapeutic decisions.

The aim of the study is to fill the evidence gap regarding the diagnostic and prognostic value of biomarkers, as well as the type and burden of arrhythmias in patients with myocarditis.

This will be a non-interventional, observational study. The study will include 100 adult patients with confirmed (based on clinical findings, in accordance with applicable guidelines) first myocarditis episode, who agree to participate in the study.

During the multicenter observational study will be collected basic demographic data, current diagnosis, current disease history and clinical presentation of symptoms, laboratory tests results and all other additional tests carried out during or after index hospitalization. During the index hospitalization peripheral venous blood (10 ml) will be collected to obtain serum for further diagnostic tests (i.e. biochemical, genetic). The obtained material will be stored frozen until analysis. The tested biomarkers will include those that have a confirmed role in the diagnosis of myocardial necrosis, in inflammatory processes and fibrosis of the myocardium, participate in the pathophysiology of arrhythmia and heart failure development, i.e. high sensitive troponin, N-terminal-pro Brain Natriuretic Peptide (NT-proBNP), Galectin-3, (Suppression of Tumorigenicity 2) ST2.

Additionally, in selected cases, when a biopsy of the heart is performed in the course of the independent diagnostic procedure, the heart muscle biopsies will be analyzed. In the collected material (both in blood and biopsy samples) immunohistochemistry, virology and genetic research will be performed for specific antibodies and genetic material of pathogens causing myocarditis (mainly viruses, i.e. parvovirus B19, coxsackie, adenovirus).

The immunogenetic predisposition, as well as gene profiling of people who have become ill with myocarditis will also be sought.

In addition, patients will undergo prolonged ECG Holter monitoring for up to 7 days from the moment of consenting to participate in the study. Registered ECG recordings will be evaluated after the completed follow-up period. Then, after 3-months form inclusion in the study, a control visit will be made assessing the clinical condition of patients, clinical examination, collection of blood samples, standard resting 12-lead ECG, and 7-day ECG-Holter monitoring. Other study endpoints will be assessed after 1-year observation. The next stage will be the analysis of clinical history, obtained results of ECG monitoring, biomarkers and additional tests.

ELIGIBILITY:
Inclusion Criteria:

* clinically suspected myocarditis
* age ≥ 18 years
* signed informed consent to participate in the study

Exclusion Criteria:

* previous history of heart failure
* already Implanted implantable cardioverter-defibrillator (ICD), cardiac resynchronization therapy (CRT) or pacemaker (PM)
* history of percutaneous ablation due to arrhythmias
* history of arrhythmias or conduction disorders
* active cancer
* advanced chronic kidney disease
* chronic inflammatory disease
* previous or current myocardial infarction
* current myocardial ischemia as the cause of arrhythmia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients admitted to the hospital having clinically suspected myocarditis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of type and burden of arrhythmia using Holter-ECG monitoring in patients with myocarditis. | 3 months
  During the Holter-ECG monitoring type and burden of arrhythmias or cardiac rhythm disorders will be assessed.
Time to occurrence of new heart failure, heart failure hospitalizations or heart failure outpatient visits. | 1 year
  it will be assessed on clinical interview during control visits
Time to occurrence of cardiovascular hospitalization. | 1 year
  it will be assessed on clinical interview during control visits
Time to occurrence to left ventricular systolic dysfunction. | 1 year
  left ventricular systolic dysfunction occurrence will be assessed using echocardiography during control visits.
Time to occurrence to left ventricular diastolic dysfunction. | 1 year
  left ventricular diastolic dysfunction occurrence will be assessed using echocardiography during control visits.

SECONDARY OUTCOMES:
Correlation of serum biomarkers concentrations with cardiac remodeling | 1 year
Correlation of serum biomarkers concentrations with inflammation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Grzegorz Opolski, Professor, Study Chair — Medical University of Warsaw; Krzysztof J Filipiak, Professor, Study Chair — Medical University of Warsaw
Locations (1):
- 1st Chair and Department of Cardiology, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
after contact
Supporting Information: Study Protocol, ICF
Access Criteria: principal investigator approval